CLINICAL TRIAL: NCT06012929
Title: A Pilot Study, Open-Label Study of ONC201 for Refractory Meningioma
Brief Title: A Study of ONC201 for Refractory Meningioma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Protocol not moving forward.
Sponsor: University of Nebraska (Other)
Collaborators: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0137-24-FB
Record Dates: First submitted 2023-08-03; First posted 2023-08-28 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-01

CONDITIONS: Meningioma; Refractory Meningioma; Relapsed Meningioma
MeSH Terms: conditions — Meningioma | interventions — TIC10 compound

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I - Presurgical (Experimental): Participants who will be undergoing surgery to remove their meningioma will receive two doses of ONC201 prior to their surgery. ONC201 is taken by mouth at 625 mg per dose. ONC201 will be taken once per week with the second dose taken approximately 24 hours prior to surgery.
  Interventions: Drug: ONC201
- Arm II - ONC201 treatment only (Experimental): Participants will receive one dose of ONC201 per week until progression. ONC201 is taken by mouth at 625 mg per dose.
  Interventions: Drug: ONC201

INTERVENTIONS:
Drug: ONC201 — ONC201 is an oral medication given once per week
  Other Names: dordaviprone

SUMMARY:
The goal of this clinical trial is to learn about treatment for a type of brain tumor called a meningioma. This study will enroll two groups of people. One group will be for people who will receive surgery to remove their brain tumor. The other group will be for people who have previously received treatment for their brain tumor but do not have any other available options for treatment.

The primary goals of this study are:

1. To measure how much of the study drug is present in tumor tissue taken from patients during surgery to remove their brain tumor
2. To measure the length of time between a study participant's first dose of study treatment until the time when their brain tumor gets worse or their death

DETAILED DESCRIPTION:
Patients will be enrolled in one of two arms, either the presurgical arm or the treatment arm. Patients who will be undergoing surgery to remove their meningioma will be enrolled to Arm I. Patients who have previously received treatment for their meningioma but have exhausted all reasonable treatment options will be enrolled to Arm II.

All patients will take the study medication, ONC201, by mouth once per week at a dose of 625 mg.

* Arm I patients will receive two doses of ONC201 prior to surgery, with the second dose occurring approximately 24 hours before surgery.
* Arm II patients will receive one 625 mg dose of ONC201 per week until disease progression or intolerable toxicity.

Primary Objectives

1. To evaluate the concentration of ONC201 in resected meningioma tissue (Arm I)
2. To measure progression-free survival in patients receiving ONC201 who have exhausted all other reasonable treatment options (Arm II)

Secondary Objectives

1. To evaluate tumor response via radiographic imaging following treatment with ONC201
2. To correlate dopamine receptor D2 (DRD2) expression with tumor response to treatment via molecular studies performed on archival and fresh tissue
3. To determine overall survival
4. To determine the efficacy of adding bevacizumab to ONC201 in patients who have progressed on ONC201 alone

ELIGIBILITY:
Inclusion Criteria:

For both study arms:

1. Brain imaging demonstrating a meningioma for which resection has been recommended (Arm I) or any subject with pathologically proven meningioma without reasonable surgical options for complete resection, or reasonable radiation therapy options, determined by neurosurgery and radiation oncology opinions (Arm II)
2. Age > 18 years old at time of study entry (consent) or adult male or female (For Nebraska, age of consent is ≥19 years old)
3. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
4. Adequate organ and marrow function as defined below:

   1. Absolute neutrophil count ≥1,000/mm3 without growth factor use ≤ 7 days prior to treatment (cycle 1 day 1, C1D1)
   2. Hemoglobin >8.0 mg/dL without red blood cell transfusion ≤ 3 days prior to C1D1
   3. Total serum bilirubin <1.5 X upper limit of normal (ULN), except in cases of Gilbert's disease
   4. Aspartate aminotransferase (AST) (SGOT)/Alanine transaminase (ALT) (SGPT) ≤2 X ULN secondary to tumor
   5. Serum creatinine ≤ 1.5 X ULN (OR creatinine clearance ≥ 60 mL/min/1.73 m2)
5. Ability to understand and the willingness to sign a written informed consent document.
6. Female subjects must be surgically sterile or be postmenopausal, or must agree to use effective contraception while on ONC201 and for at least 90 days after completion of treatment. Male subjects must be surgically sterile or must agree to use effective contraception while on ONC201 and for at least 90 days after completion of treatment. The decision of effective contraception will be based on the judgment of the principal investigator or a designated associate.
7. Any number of prior medical therapies is allowed but not required.
8. Multifocal disease is allowed.
9. Subjects with history of neurofibromatosis may have other stable central nervous system (CNS) tumors (schwannoma, acoustic neuroma or ependymoma) if lesions have been stable for 6 months.

   For Arm II only:
10. Progression by Macdonald criteria: increase in size of the measurable primary lesion on imaging by 25% or more (bidirectional area). Progressive disease must based on scans done within 12 months or fewer of each other.
11. Subject must have no reasonable surgical or radiation therapy options, determined by neurosurgery and radiation oncology opinions.
12. Evidence of progressive disease at least 24 weeks after completion of radiation (external beam, interstitial brachytherapy, or radiosurgery).
13. Subject who elected to have partial tumor resection after confirmed progressive disease may still be considered, but radiographic measurable residual tumor(s) are required at baseline
14. Stable or decreasing steroid dose for two weeks.
15. Archival tissue must be available for correlative studies-a minimum of ten slides to be eligible, with up to 20 slides requested.

Exclusion Criteria:

1. Participation in another clinical study with an investigational product during the last 28 days.
2. Active chemotherapy, including other investigational agents within 28 days of study treatment.
3. Craniotomy or other major surgery within 28 days of registration.
4. Evidence of metastatic meningiomas (as defined by extracranial meningiomas).
5. Known active bacterial, fungal or viral infection including hepatitis B (HBV), hepatitis C (HCV).
6. Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness.
7. Any of the following in the previous 6 months: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, or cerebrovascular accident. Subjects planning to continue on study after progression with the addition of bevacizumab cannot have uncontrolled hypertension, nephrotic syndrome, or had a history of intracranial bleeding or GI hemorrhage in the last 6 months.
8. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, or in the judgment of the investigator would make the subject inappropriate for entry into the study.
9. Concomitant treatment with strong inhibitors of cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4) inhibitors or inducers. Subject must discontinue the drug for 14 days prior to registration.
10. Prolongation of QT/corrected QT interval by Fridericia (QT/QTcF) interval (QTc interval >480 milliseconds) using Frederica's QT correction formula on two ECGs separated by at least 48 hours.
11. A history of Torsades de pointes or heart failure, hypokalemia, or family history of prolonged QT Syndrome.
12. Concomitant use of medication(s) known to prolong the QT/QTc interval.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2026-12 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Evaluation of ONC201 concentration in resected meningioma tissue | Up to 12 months
  Tumor tissue will be collected from Arm I participants at the time of surgical resection. The samples will be analyzed for the concentration of ONC201 in the tissue.
Evaluation of progression-free survival (PFS) | Up to 18 months
  PFS at 6 months will be evaluated in participants assigned to Arm II. PFS is defined as the time from the start of study treatment to the time of disease progression or death. Participants without progression and who are alive at the time of last follow-up will be censored.

SECONDARY OUTCOMES:
Evaluation of tumor response from ONC201 on imaging | Up to 24 months
  Tumor response from ONC201 on imaging will be measured by contrast-enhanced brain MRI completed every 12 weeks. Response will be determined using Macdonald criteria. The Macdonald criteria evaluates the status of lesions present on baseline imaging, the appearance of new lesions, corticosteroid use, and clinical status to determine the appropriate response category. The possible response categories include complete response, partial response, stable disease, and progressive disease.
Correlation of DRD2 expression with tumor response | Up to 12 months
  Archival formalin-fixed paraffin embedded (FFPE) tumor tissue samples will be collected from Arm II participants at the time of study enrollment. The tissue samples will be tested for the level of DRD2 expression. The mechanism of action for the study medication, ONC201, is the through the inhibition of DRD2 receptors, a type of dopamine receptor. DRD2 expression will subsequently be correlated with best response and compared by response categories with Kruskal-Wallis test or Wilcoxon rank sum test, depending on the number of response levels.
Evaluation of the efficacy of adding bevacizumab to ONC201 following disease progression | Up to 24 months
  Tumor response from ONC201 with bevacizumab on imaging will be measured by contrast-enhanced brain MRI completed every 12 weeks. Response will be determined using Macdonald criteria. The Macdonald criteria evaluates the status of lesions present on baseline imaging, the appearance of new lesions, corticosteroid use, and clinical status to determine the appropriate response category. The possible response categories include complete response, partial response, stable disease, and progressive disease.

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Shonka, MD, Principal Investigator — University of Nebraska

IPD SHARING:
Plan to Share IPD: No